CLINICAL TRIAL: NCT01689129
Title: A 6-Month, Multicenter, Randomized, Open-label, Parallel-group Study Comparing the Efficacy and Safety of a New Formulation of Insulin Glargine and Lantus® in Japanese Patients With Type 1 Diabetes Mellitus With a 6-month Safety Extension Period
Brief Title: Comparison of a New Formulation of Insulin Glargine With Lantus® in Japanese Patients With Type 1 Diabetes Mellitus
Acronym: EDITION JP I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12449; U1111-1130-3513 (Other: UTN)
Record Dates: First submitted 2012-09-14; First posted 2012-09-21 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New formulation of insulin glargine (Experimental): once daily in the evening on-top of mealtime insulin
  Interventions: Drug: Insulin glargine new formulation (HOE901)
- Lantus (insulin glargine) (Active Comparator): once daily in the evening on-top of mealtime insulin
  Interventions: Drug: Insulin glargine (HOE901) (Lantus)

INTERVENTIONS:
Drug: Insulin glargine new formulation (HOE901) — Pharmaceutical form: solution Route of administration: subcutaneous
  Arms: New formulation of insulin glargine
Drug: Insulin glargine (HOE901) (Lantus) — Pharmaceutical form: solution Route of administration: subcutaneous
  Other Names: Lantus
  Arms: Lantus (insulin glargine)

SUMMARY:
Primary Objective:

To compare the efficacy of a new formulation of insulin glargine and Lantus in terms of change of HbA1c from baseline to endpoint (scheduled at month 6 [week 26]) in japanese patients with type 1 diabetes mellitus

Secondary Objectives:

To compare a new formulation of insulin glargine and Lantus in terms of change in fasting plasma glucose (FPG), preinjection plasma glucose, 8-point self-measured plasma glucose (SMPG) profile.

To compare a new formulation of insulin glargine and Lantus in terms of occurrence of hypoglycemia

DETAILED DESCRIPTION:
The duration of study will consist of:

* Up to 2-week screening period;
* 6-month open-label comparative efficacy and safety treatment period;
* 6-month open-label comparative safety extension period;
* 4-week post-treatment safety follow-up period

ELIGIBILITY:
Inclusion criteria:

* Patients with type 1 diabetes mellitus

Exclusion criteria:

* Age < 18 years at screening visit;
* HbA1c < 7.0 % or > 10.0 % (national glycohemoglobin standardization program [NGSP] value) at screening visit;
* Patients less than 1 year before screening visit on any basal plus mealtime insulin;
* Patients not on stable insulin dose (±20% total basal insulin dose) in the last 30 days prior to screening visit;
* Patients using pre-mix insulins, human regular insulin as mealtime insulin and/or any glucose-lowering drugs other than basal insulin and mealtime rapid-insulin analogue in the last 3 months before screening visit;
* Use of an insulin pump in the last 6 months before screening visit and/or plan to switch to insulin pump in next 12 months;
* Severe hypoglycemia resulting in coma/seizures, and/or hospitalization for diabetic ketoacidosis in the last 6 months before screening visit;
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require treatment (eq, laser, surgical treatment or injectable drugs) during the study period.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | baseline, 6 months

SECONDARY OUTCOMES:
Percentage of HbA1c responders (HbA1c < 7%; < 6.5%) | up to 6 months
Change from baseline in FPG | baseline, 6 months
Change from baseline in pre-basal insulin injection SMPG | baseline, 6 months
Change from baseline in 8-point SMPG profiles | baseline, 6 months
Change from baseline in 24-hour mean plasma glucose of SMPG profiles (mean of 8-point values) | baseline, 6 months
Change from baseline in variability of plasma glucose profile | baseline, 6 months
Change from baseline in daily basal insulin dose | baseline, 6 months
Number of Patients with various types of Hypoglycemia Events | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (22):
- Japan (22):
  - Investigational Site Number 392119, Amagasaki-Shi
  - Investigational Site Number 392106, Chūōku
  - Investigational Site Number 392107, Chūōku
  - Investigational Site Number 392110, Ebina-Shi
  - Investigational Site Number 392115, Higashiosaka-Shi
  - Investigational Site Number 392117, Izumisano
  - Investigational Site Number 392109, Kamakura-Shi
  - Investigational Site Number 392101, Koriyama-Shi
  - Investigational Site Number 392121, Kurashiki-Shi
  - Investigational Site Number 392112, Nagoya
  - Investigational Site Number 392120, Nishinomiya-Shi
  - Investigational Site Number 392113, Osaka
  - Investigational Site Number 392116, Osaka
  - Investigational Site Number 392118, Osaka
  - Investigational Site Number 392104, Shinjuku-Ku
  - Investigational Site Number 392105, Shinjuku-Ku
  - Investigational Site Number 392111, Shizuoka
  - Investigational Site Number 392114, Takatsuki-Shi
  - Investigational Site Number 392122, Tokushima
  - Investigational Site Number 392103, Tomioka-Shi
  - Investigational Site Number 392102, Ushiku-Shi
  - Investigational Site Number 392108, Yokohama

REFERENCES:
- [Derived] Matsuhisa M, Koyama M, Cheng X, Takahashi Y, Riddle MC, Bolli GB, Hirose T; EDITION JP 1 study group. New insulin glargine 300 U/ml versus glargine 100 U/ml in Japanese adults with type 1 diabetes using basal and mealtime insulin: glucose control and hypoglycaemia in a randomized controlled trial (EDITION JP 1). Diabetes Obes Metab. 2016 Apr;18(4):375-83. doi: 10.1111/dom.12619. Epub 2016 Feb 1. PMID 26662964